CLINICAL TRIAL: NCT02119806
Title: Decreasing the Incidence of Delirium After Cardiac Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jacques Neelankavil, HS Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Delirium 13-001412
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: C.Surgical Procedure; Cardiac; Delirium
Keywords: cardiac surgery, benzodiazepines, delirium
MeSH Terms: conditions — Delirium | interventions — Benzodiazepines; Midazolam; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benzodiazepine group (Active Comparator): 1. Premedication 0.02mg/kg-0.1mg/kg of Benzodiazepine ;
  2. Maintenance 0.8 minimum alveolar concentration of inhaled anesthetic (MAC) and 10-30mcg/kg of fentanyl;
  3. Postoperative 10-100mcg/kg/min of propofol
  Interventions: Drug: Benzodiazepine; Drug: Fentanyl; Drug: Propofol
- Non-benzodiazepine group (Active Comparator): 1. Premedication 0-50mg of propofol and/or 0-250mcg of fentanyl;
  2. Maintenance 0.8 minimum alveolar concentration of inhaled anesthetic (MAC) and 10-30mcg/kg of fentanyl;
  3. Postoperative 10-100mcg/kg/min of propofol
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Benzodiazepine — Receive as premedication in the Benzodiazepine group.
  Other Names: Midazolam; Versed
  Arms: Benzodiazepine group
Drug: Fentanyl — Receive as maintenance in the Benzodiazepine group. Can receive as premedication in the Non-Benzodiazepine group. Receive as maintenance in the Non-Benzodiazepine group.
  Other Names: Fentanil
Drug: Propofol — Receive postoperatively in the Benzodiazepine group. Can receive as premedication in the Non-Benzodiazepine group. Receive postoperatively in the Non-Can receive as premedication in the Non-Benzodiazepine group.
  Other Names: Diprivan

SUMMARY:
In critically ill surgical patients, delirium (confusion and disorientation) is extremely common and is associated with longer hospital length of stay, mortality, cost, and long term cognitive impairment. The goal of the study is to establish whether benzodiazepines (a sedative, anti-anxiety drug) should be used as part of standard of care or be eliminated by comparing the chances of delirium in cardiac surgery patients between two groups: a group that receives benzodiazepines during surgery versus a group that does not receive benzodiazepines during surgery. Benzodiazepines have historically been used in cardiac anesthesia to decrease the risk of anesthesia awareness. The current standard of care is to keep the patient on inhaled anesthesia throughout the surgery which eliminates the need for intraoperative use of benzodiazepines. Benzodiazepines are still used based on practitioner preference. Findings of this study will allow all anesthesiologists to make more informed decisions about what level of care our patients need.

DETAILED DESCRIPTION:
In critically ill surgical patients, delirium is extremely common and is associated with longer hospital length of stay, mortality, cost, and long term cognitive impairment. Benzodiazepine usage is common in anesthetic practice, and ICU literature demonstrates that limiting post-operative benzodiazepines decreases the incidence of delirium. However, the avoidance of preoperative and intraoperative benzodiazepines during cardiac surgery has not been studied in terms of its effect on delirium. The goal of the study is establish whether benzodiazepines should be used as part of standard of care or be eliminated by comparing the incidence of delirium in cardiac surgical patients when randomized to a group that receives benzodiazepines versus a group that does not receive benzodiazepines.

Potential subjects will be identified and recruited the day before surgery by primary investigators. Patients undergoing coronary artery bypass grafting or single valve procedures that consent to participate will be enrolled in the study. These patients may be consented during the pre-operative period. Patients will be informed that whether they enroll in the study or not, they will be receiving standard clinical care. Only subjects meeting all inclusion criteria and requirements for continuation in the study will be consented.

Patient will be randomized by age (age is a predictor of delirium) to 3 groups:

* >80 years of age;
* 70-80 years of age;
* < 70 years of age.

Within these 3 groups, patients will be randomized to receive benzodiazepines during cardiac surgery or not. The anesthesiologist in the operating room will not be blinded to the group; however, the intensive care physician evaluating for delirium will be blinded to the treatment groups.

Benzodiazepine group:

1. Premedication 0.02mg/kg-0.1mg/kg of midazolam;
2. Maintenance 0.8 minimum alveolar concentration of inhaled anesthetic (MAC) and 10-30mcg/kg of fentanyl;
3. Postoperative 10-100mcg/kg/min of propofol

Non-benzodiazepine group:

1. Premedication 0-50mg of propofol and/or 0-250mcg of fentanyl;
2. Maintenance 0.8 minimum alveolar concentration of inhaled anesthetic (MAC) and 10-30mcg/kg of fentanyl;
3. Postoperative 10-100mcg/kg/min of propofol

Delirium can now be reliably diagnosed by non-psychiatrists in critically ill patients in less than 2 minutes through the use of validated monitoring instruments such as the Confusion Assessment Method for the ICU (CAM-ICU).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients' undergoing coronary artery bypass grafting or single valve procedures.

Exclusion Criteria:

* Patients who have baseline cognitive dysfunction,
* Patients with hearing problems,
* Patients currently on benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Delirium | less than 2 minutes
  Delirium can now be reliably diagnosed by non-psychiatrists in critically ill patients in less than 2 minutes through the use of validated monitoring instruments such as the Confusion Assessment Method for the ICU (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Neelankavil, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology, Los Angeles, California, United States

REFERENCES:
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Girard TD, Jackson JC, Pandharipande PP, Pun BT, Thompson JL, Shintani AK, Gordon SM, Canonico AE, Dittus RS, Bernard GR, Ely EW. Delirium as a predictor of long-term cognitive impairment in survivors of critical illness. Crit Care Med. 2010 Jul;38(7):1513-20. doi: 10.1097/CCM.0b013e3181e47be1. PMID 20473145
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384